CLINICAL TRIAL: NCT01922440
Title: PARADIGHM (Physicians Advancing Disease Knowledge in Hypoparathyroidism): A Registry for Patients With Chronic Hypoparathyroidism
Brief Title: A Registry for Participants With Chronic Hypoparathyroidism
Acronym: PARADIGHM
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PAR-R13-001; EUPAS16927 (Other: ENCePP EU PAS)
Record Dates: First submitted 2013-08-01; First posted 2013-08-14 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hypoparathyroidism
Keywords: Chronic Hypoparathyroidism; rhPTH(1-84); Observational study; parathyroid hormone (PTH); Drug registry; rhPTH(1-34)
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Natpar(a): Participants receiving parathyroid hormone (rhPTH(1-84) (Natpar[a]) for treatment of chronic hypoparathyroidism as per standard clinical practice will be enrolled and evaluated during the study period.
  Interventions: Other: No intervention
- Conventional Therapy: Participants receiving conventional therapy/standard of care (including calcium supplements, active vitamin D, vitamin D) for treatment of chronic hypoparathyroidism as per standard clinical practice will be enrolled and evaluated during the study period.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to find out the long-term safety and effectiveness profile of recombinant human parathyroid hormone (1-84) (rhPTH[1-84]) treatment in participants with chronic hypoparathyroidism under conditions of routine clinical practice.

Participants will be treated according to their clinic's standard practice determined by the treating doctors. Each participant will fill out a study questionnaire during a routine doctor visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with chronic hypoparathyroidism, that is, hypoparathyroidism with a duration of longer than 6 months, including:

  1. Adult participants (greater than or equal to [>=] 18 years of age) who are receiving for chronic hypoparathyroidism any of the following options: standard therapy, standard therapy plus rhPTH(1-84), or rhPTH(1-84) therapy alone.
  2. Pediatric participants (less than [<] 18 years of age) who are receiving for chronic hypoparathyroidism any of the following options: standard therapy, standard therapy plus rhPTH(1-84), or rhPTH(1-84) therapy alone.

Exclusion Criteria:

* Participants or legally acceptable representatives unable to provide informed consent.
* Participants using rhPTH(1-34) or who used rhPTH(1-34) for more than 2 years are excluded. Participants who had been treated with rhPTH(1-34) within 3 months of enrollment are also excluded as are participants currently using rhPTH(1-34).

FOR US SITES ONLY: Participants treated with rhPTH(1-84) prior to the US recall may use rhPTH(1-34) only while rhPTH(1-84) is unavailable due to the recall.

* Participants currently enrolled in an interventional clinical study (whether or not the study is related to hypoparathyroidism); note that this does not include participants enrolled in other observational registries.
* History of hypoparathyroidism resulting from impaired responsiveness to PTH (pseudohypoparathyroidism).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This global registry is expected to enroll a minimum of 900 participants, of whom at least 300 will be participants treated with rhPTH(1-84) and at least 600 will be participants receiving standard of care. Protocol amendment 9 revised the sample size: up to 164 additional participants treated with rhPTH(1-84) (ie, up to a total of 464 participants in that cohort) will be enrolled as needed to ensure the availability of 104 rhPTH(1-84)-treated participants with a full 10 years of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1339 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2034-11-30 (Estimated); Study Completion 2034-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 24-Hour Urine Calcium | Baseline up to 10 years (follow-up)
  Change from baseline in 24-hour urine calcium will be evaluated.
Change from Baseline in Serum Calcium | Baseline up to 10 years (follow-up)
  Change from baseline in serum calcium will be evaluated.
Change from Baseline in Serum Albumin | Baseline up to 10 years (follow-up)
  Change from baseline in serum albumin will be evaluated.
Change from Baseline in Albumin-Corrected Total Calcium | Baseline up to 10 years (follow-up)
  Change from baseline in albumin-corrected total calcium will be evaluated.
Change from Baseline in Serum Ionized Calcium | Baseline up to 10 years (follow-up)
  Change from baseline in serum ionized calcium will be evaluated.
Change from Baseline in Serum Magnesium | Baseline up to 10 years (follow-up)
  Change from baseline in serum magnesium will be evaluated.
Change from Baseline in Serum Phosphate | Baseline up to 10 years (follow-up)
  Change from baseline in serum phosphate will be evaluated
Change from Baseline in 25-Hydroxy (25-OH) Vitamin D results | Baseline up to 10 years (follow-up)
  Change from baseline in 25-OH vitamin D will be evaluated.
Change from Baseline in Serum Creatinine | Baseline up to 10 years (follow-up)
  Change from baseline in serum creatinine will be evaluated.
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR; calculated) | Baseline up to 10 years (follow-up)
  Change from baseline in eGFR; calculated will be evaluated.
Change from Baseline in 24-Hour Urine Protein | Baseline up to 10 years (follow-up)
  Change from Baseline in 24-hour urine protein will be evaluated.
Incidence Rate of the Renal Events | Baseline up to 10 years (follow-up)
  Incidence rate of the renal events will be recorded for nephrolithiasis, nephrocalcinosis, hospitalization/emergency room visits for renal events.
Incidence Rate of the Soft Tissue Calcifications (site) | Baseline up to 10 years (follow-up)
  Incidence rate of the soft tissue calcifications (site) will be recorded.
Incidence Rate of the Cataract | Baseline up to 10 years (follow-up)
  Incidence rate of the cataract will be recorded by questionnaire (present/not present).
Incidence Rate of the Bone Fractures (site) | Baseline up to 10 years (follow-up)
  Incidence rate of the bone fractures (site) will be recorded.
Incidence Rate of the Cardiovascular Events | Baseline up to 10 years (follow-up)
  Incidence rate of the cardiovascular events will be calculated for this clinical outcome. Cardiovascular events include myocardial infarction, stroke, arrhythmia.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 10 years (follow-up)
  An AE is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product. An SAE is any untoward medical occurrence (whether considered to be related to study product or not) that at any dose results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality or birth defect, an important medical event.

SECONDARY OUTCOMES:
Health-related Quality of Life (HRQoL) | Baseline up to 10 years (follow-up)
  Health-Related Quality of Life (HRQoL), as measured by the short-form-10 (SF-10) for pediatrics, short-form-36 (SF-36) for adults will be examined longitudinally using methods for continuous data.
Disease-specific Patient-reported Outcome Measures | Baseline up to 10 years (follow-up)
  Chronic hypoparathyroidism patient-reported outcome will be recorded as measured by the hypoparathyroidism multi-symptom diary (HPT-SD).
Rate of Hospitalization/Emergency Room (ER) Visits | Baseline up to 10 years (follow-up)
  The rate of hospitalizations and ER visits during follow-up will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (100):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Medical Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Dr. Joselito Cabaccan, San Jose, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Thyroid & Endocrine Center of Florida, Sarasota, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Suburban Endocrinology & Diabetes, Arlington Heights, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Tilak Mallik, MD F.A.C.E., LCC, Marrero, Louisiana
  - Model Clinical Research, Baltimore, Maryland
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Diabetes & Endocrine Associates, Methodist Physicians Clinic Diabetes and Endocrine Specialists, Omaha, Nebraska
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Northern Nevada Endocrinology, Reno, Nevada
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Med Endocrine Specialists, Albany, New York
  - Brokhin Medical PC, Brooklyn, New York
  - Gerald Friedman Diabetes Institute, New York, New York
  - Columbia University Medical Center, New York, New York
  - Endocrine Associates of Long Island, P.C., Smithtown, New York
  - University Physicians Group Research Division, Staten Island, New York
  - State University Of New York Upstate Medical University, Syracuse, New York
  - Mecklenburg Medical Group, Charlotte, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Endocrinology Associates of Armstrong, Indiana, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - Hallett Center for Diabetes and Endocrinology, East Providence, Rhode Island
  - University of South Carolina, Columbia, South Carolina
  - Texas Diabetes and Endocrinology, P.A., Austin, Texas
  - Thyroid Endocrinology and Diabetes, Dallas, Texas
  - Academy of Diabetes Thyroid and Endocrine, El Paso, Texas
  - Diabetes and Thyroid Center of Fort Worth, PLLC, Fort Worth, Texas
  - University of Vermont, South Burlington, Vermont
  - University of Wisconsin, Madison, Wisconsin
- Austria (2):
  - Medizinische Universitaetsklinik Graz, Universitätsklinik Für Innere Medizin Graz, Graz
  - AKH Wien, Universitaetsklinik fuer Innere Medizin III, Vienna
- Canada (2):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University, Oakville, Ontario
- Denmark (4):
  - Aallborg University Hospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Nordsjaellands Hospital - Hillerod, Hilleroed
  - Regions Hospitalet Viborg, Viborg
- Germany (17):
  - Diakonie-Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - University of Leipzig, Leipzig, Saxony
  - Universitaetsklinik Aachen, Aachen
  - Charite-Universitiitsmedizin Berlin (CCM), Berlin
  - Praxis an der Kaiserreiche, Berlin
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Endokrinologikum Frankfurt, Frankfurt
  - MVZ endokrinologikum Göttingen, Göttingen
  - Universitaet Zur Luebeck, Lübeck
  - Medicover Neuroendokrinologie MVZ, München
  - Medicover Neu-Ulm Mvz, Neu-Ulm
  - Medicover Oldenburg MVZ, Oldenburg
  - Medicover Saarbuecken Mvz, Saarbrücken
  - Endokrinologie Zentrum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (5):
  - General Hospital Of Athens - Korgialenio-Benakio E.E.S., Athens
  - General Hospital of Athens Georgios Gennimatas, Athens
  - General Hospital of Athens Alexandra, Athens
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Hippokrateion General Hospital of Thessaloniki, Thessaloniki
- Italy (4):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza - Ospedale Molinette, Torino
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Spesialistsentret Pilestredet Park, Oslo
- Spain (3):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (4):
  - Universitetssjukhuset I Linkoping, Linköping
  - Universitetssjukhuset I Orebro, Örebro
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Akademiska Sjukhuset - Uppsala University Hospital, Uppsala
- United Kingdom (3):
  - Queen Elizabeth Hospital-Mindelsohn Way, Birmingham, England
  - University of Hospitals of Leicester, Leicester
  - Norfolk And Norwich University Hospital - Norwich Medical School, Norwich

REFERENCES:
- [Derived] Gittoes N, Rejnmark L, Ing SW, Brandi ML, Bjornsdottir S, Hahner S, Hofbauer LC, Houillier P, Khan AA, Levine MA, Mannstadt M, Shoback DM, Vokes TJ, Zhang P, Marelli C, Germak J, Clarke BL. The PARADIGHM (physicians advancing disease knowledge in hypoparathyroidism) registry for patients with chronic hypoparathyroidism: study protocol and interim baseline patient characteristics. BMC Endocr Disord. 2021 Nov 20;21(1):232. doi: 10.1186/s12902-021-00888-2. PMID 34801015
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd14db2bf003ab46a03